CLINICAL TRIAL: NCT03525977
Title: Impact of Fascia Iliaca Block on Pain Outcomes and Opioid Consumption for Hip Fracture Patients-A Prospective, Randomized Study
Brief Title: Impact of Fascia Iliaca Block in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Mai P. Nguyen, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E18046
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Hip Fractures (i.e. Femoral Neck or Intertrochanteric Hip Fractures)
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control arm will receive pain control via traditional oral and intravenous pain medications such as opioids and non-steroidal anti-inflammatory medication as needed.
- Fascia iliaca block (Experimental): Patients in the intervention arm will receive the regional fascia iliaca block performed by the anesthesiologists on call.
  Interventions: Procedure: Fascia iliaca block arm

INTERVENTIONS:
Procedure: Fascia iliaca block arm — The fascia iliaca block will be performed by the anesthesiologist on call
  Other Names: FIB
  Arms: Fascia iliaca block

SUMMARY:
The study is a prospective randomized examining the impact of fascia iliaca block on perioperative pain control and post operative ambulation in patients with hip fractures.

DETAILED DESCRIPTION:
Regional anesthesia is an important element of multimodal pain control regimen for surgical patients. Recently, regional anesthesia using a fascia iliaca block (FIB) to help treat pain in patients who present with hip fractures has been gaining popularity and has been incorporated as part of a multi-modal pain control protocol in many centers. It is commonly offered in addition to oral and intravenous medications to help patients deal with pain in the perioperative period. The block is done by an anesthesiologist under anesthesia using ultrasound guidance. We propose a prospective, randomized study evaluating the efficacy of the FIB as an adjunct in the pre-operative or postoperative period for pain control as measured by visual analog scale (VAS) scores and morphine equivalent dosing (MED), as well as its efficacy in promoting patient participation in physical therapy postoperatively in patients who present with hip fractures. We hypothesize that those patients who receive FIBs will report lower VAS scores as well as decreased narcotic requirement at all time points; and have improved participation in therapy when measured by ambulation distance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with femoral neck and intertrochanteric hip fractures
* At least 18 years of age
* Require operative management

Exclusion Criteria:

* Poly-trauma patients
* Pathologic fractures
* Patient who required revision procedures
* Patients with chronic opioid use
* Patients with a clinical status that precludes verbal pain assessment such as dementia, head injuries, and unwillingness to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Pain level | Pre operatively
  Visual analog scale scores (from 0-10 with 0 being no pain and 10 being the worst pain)
Pain medication requirement | Pre operatively
  Morphine equivalent dosing
Pain level | Four hours after surgery
  Visual analog scale scores (from 0-10 with 0 being no pain and 10 being the worst pain)
Pain medication requirement | Four hours after surgery
  Morphine equivalent dosing
Pain level | One day after surgery
  Visual analog scale scores (from 0-10 with 0 being no pain and 10 being the worst pain)
Pain medication requirement | One day after surgery
  Morphine equivalent dosing
Pain level | Two days after surgery
  Visual analog scale scores (from 0-10 with 0 being no pain and 10 being the worst pain)
Pain medication requirement | Two days after surgery
  Morphine equivalent dosing
Pain level | Three days after surgery
  Visual analog scale scores and morphine equivalent dosing
Pain medication requirement | Three days after surgery
  Morphine equivalent dosing

SECONDARY OUTCOMES:
Ambulation distance | Two days after surgery
  Ambulation distance with physical therapy post op

CONTACTS AND LOCATIONS:
Overall Officials: Mai Nguyen, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- University Medical Center, El Paso, Texas, United States

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043